CLINICAL TRIAL: NCT05525741
Title: Assessment of Circulating Fubctional Mitochondrias in Vitiligo Patients as Compared to Controls
Brief Title: Assessment of Circulating Fubctional Mitochondrias in Vitiligo Patients
Acronym: MFC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 22-PP-10
Record Dates: First submitted 2022-08-23; First posted 2022-09-02 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Skin and Connective Tissue Diseases
MeSH Terms: conditions — Skin and Connective Tissue Diseases

STUDY DESIGN:
Intervention Model Description: Patients with non segmental vitiligo compared to healthy volunteers (1st degree family of vitiligo patients) atopic dermatitis, psoriasis and alopecia areata patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitiligo Group (Experimental): If the subject consents and they meet all the criteria a 20 ml blood sample will be taken.
  Interventions: Other: Non segmental vitiligo
- Volunteers Group (Other): If the subject consents and they meet all the criteria a 20 ml blood sample will be taken.
  Interventions: Other: Health Volunteers

INTERVENTIONS:
Other: Non segmental vitiligo — The subjects will be selected from among those presenting for the consultation or hospitalization of the Dermatology department of the CHU de Nice. All necessary information will be given to the subjects and a briefing note will be given to them. A reflection period will be left for the subjects to sign the informed consent, and if necessary, another appointment will be scheduled for the inclusion visit.
  The Investigator:
  * Inform the subject of the goals, constraints and risks of the study and obtain written consent.
  * Conduct an examination of the subject's medical history Will verify that the subject meets all inclusion criteria and does not present any of the criteria for not including.
  If the subject consents and they meet all the criteria a 20 ml blood sample will be taken.
  Arms: Vitiligo Group
Other: Health Volunteers — The subjects will be selected from among those presenting for the consultation or hospitalization of the Dermatology department of the CHU de Nice. The family control subjects will be recruited from the vitiligos patients coming into our department. All necessary information will be given to the subjects and a briefing note will be given to them. A reflection period will be left for the subjects to sign the informed consent, and if necessary, another appointment will be scheduled for the inclusion visit.
  The Investigator:
  * Inform the subject of the goals, constraints and risks of the study and obtain written consent.
  * Conduct an examination of the subject's medical history Will verify that the subject meets all inclusion criteria and does not present any of the criteria for not including.
  If the subject consents and they meet all the criteria a 20 ml blood sample will be taken.
  Arms: Volunteers Group

SUMMARY:
To compare the level of circulating functional mitochondria in the serum of vitiligo patients as compared to controls

ELIGIBILITY:
Inclusion Criteria:

* Patients with non segmental vitiligo,
* atopic dermatitis, psoriais, alopecia areata,
* 1st degree relative of vitiligo patients.

Exclusion Criteria:

* segmental or mixed vitiligo,
* personnal history of other autoimmune disorders,
* oral use of antioxidant,
* pregant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Total number of circulating functionnal mitochondria (CFM) in the plasma | at baseline
  Level of CFM in vitiligo serum as compared to controls

SECONDARY OUTCOMES:
measuring the functionality of circulating mitochondria | At baseline
  Functional analysis of CFM in vitiligo patients as compared to controls analyzed by MFI Mito Tracker

CONTACTS AND LOCATIONS:
Overall Officials: passeron thierry, PhD, Principal Investigator — CHU de Nice, Service de Dermatologie
Locations (1):
- CHU de Nice - Hôpital de l'Archet, Nice, Alpes-maritimes, France

IPD SHARING:
Plan to Share IPD: Undecided